CLINICAL TRIAL: NCT04767126
Title: Impact of Pulmonary Rehabilitation on Peripheral Skeletal Muscle Function in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Peripheral Muscle Function in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Simone Pancera, PhD(s), Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: MAC_COPD_FDG
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Copd
Keywords: Copd; Pulmonary rehabilitation; Muscle strength
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by irreversible airway obstruction and progressive deterioration of respiratory function. Patients with COPD show a limited exercise tolerance, early fatigability and progressive dyspnea, with important consequences on the ability to sustain even mild efforts and a drastic restriction in the activities of daily living. Muscle dysfunction is a systemic manifestation of COPD that contributes to exertion intolerance in individuals with COPD to the point of compromising fundamental functional activities, such as walking. Previous studies have shown, in fact, that quadriceps strength can be reduced by 20% to 30% in patients with COPD and this value is associated with an increased risk of mortality in patients with lower strength levels. In addition, loss of muscle mass or sarcopenia also occurs with a prevalence of between 8% and 67% in patients with COPD, exacerbating the picture of muscle dysfunction.

One of the goals of respiratory rehabilitation is precisely the prevention of muscle dysfunction in patients with COPD. However, rehabilitation programs aimed at maintaining and recovering muscle strength are often lacking in guidance regarding target muscles, duration of sessions, and training intensity, while strength assessment is often limited by the timing and resources associated with the clinical setting in which it takes place. This makes it difficult to determine its short- and long-term effectiveness.

Therefore, assessment of muscle function in patients with COPD requires tests that are simple and quick to perform, but equally capable of providing quantitative data referable to a specific characteristic of muscle strength as well as indicative of the patient's overall function. In addition, complementary measurements such as body composition and muscle mass, as well as the development of predictive models and normative values of muscle function could provide additional information on the progression of muscle dysfunction in patients with COPD, allowing rehabilitation intervention to be directed toward recovery of the most compromised functions.

Therefore, the aims of this study are: 1) To evaluate the effectiveness of a standard pulmonary rehabilitation program in recovering peripheral muscle dysfunction in patients with COPD. 2) To evaluate the clinical reliability of tests commonly used to measure peripheral muscle function in the rehabilitation setting of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis (GOLD stage: II-III-IV), defined as post-bronchodilator forced expiratory volume in 1s (FEV1)/forced vital capacity < 0.7 and FEV1 < 80% predicted.

Exclusion Criteria:

* Restrictive lung disease, unstable conditions, recent exacerbation, infection, embolism, pneumothorax, thoracic or abdominal surgery (less than 3 months before recruitment).
* Cardiologic conditions like myocardial infarction (less than 6 months before recruitment), heart failure, or severe angina.
* Inability of perform the exercise training (e.g. orthopaedic conditions).
* Incapability to understand the instructions required to carry out the tests and assessments planned.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with COPD referred to the Cardiopulmonary Rehabilitation Unit of a tertiary referral sub-acute rehabilitation centre.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Lower limbs muscle power | Change from baseline through study completion, an average of 6 weeks
  Muscle power of the lower limbs measured during the sit-to-stand test
Lower limbs muscle power | Change after 3 months from study completion
  Muscle power of the lower limbs measured during the sit-to-stand test

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy

REFERENCES:
- [Background] Agusti AG. Systemic effects of chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2005;2(4):367-70; discussion 371-2. doi: 10.1513/pats.200504-026SR. PMID 16267364
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Marklund S, Bui KL, Nyberg A. Measuring and monitoring skeletal muscle function in COPD: current perspectives. Int J Chron Obstruct Pulmon Dis. 2019 Aug 19;14:1825-1838. doi: 10.2147/COPD.S178948. eCollection 2019. PMID 31695351
- [Background] Jones SE, Maddocks M, Kon SS, Canavan JL, Nolan CM, Clark AL, Polkey MI, Man WD. Sarcopenia in COPD: prevalence, clinical correlates and response to pulmonary rehabilitation. Thorax. 2015 Mar;70(3):213-8. doi: 10.1136/thoraxjnl-2014-206440. Epub 2015 Jan 5. PMID 25561517
- [Background] Nyberg A, Saey D, Maltais F. Why and How Limb Muscle Mass and Function Should Be Measured in Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2015 Sep;12(9):1269-77. doi: 10.1513/AnnalsATS.201505-278PS. PMID 26208090
- [Background] Swallow EB, Reyes D, Hopkinson NS, Man WD, Porcher R, Cetti EJ, Moore AJ, Moxham J, Polkey MI. Quadriceps strength predicts mortality in patients with moderate to severe chronic obstructive pulmonary disease. Thorax. 2007 Feb;62(2):115-20. doi: 10.1136/thx.2006.062026. Epub 2006 Nov 7. PMID 17090575